CLINICAL TRIAL: NCT04944810
Title: Bariatric, Revisional and General Surgery With Magnetic Assistance
Brief Title: Magnetic System in Bariatric and General Surgery
Status: Recruiting | Type: Observational
Sponsor: Unidad Internacional de Cirugia Bariatrica y Metabolica (Other)
Responsible Party: Principal Investigator, Guillermo Borjas, Director of the International Bariatric and Metabolic Surgery Unit, Unidad Internacional de Cirugia Bariatrica y Metabolica
Other Study IDs: UnidadInterBariatrica
Record Dates: First submitted 2021-06-10; First posted 2021-06-30 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Surgery; Bariatric Surgery Candidate
Keywords: bariatric surgery; gastric bypass; magnetic bariatric surgery; magnetic surgery; magnetic grasper; sleeve gastrectomy; revisional surgery; single-port; reduced-port

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Magnetic bariatric surgery: Perform a bariatric surgery using the magnetic device like a second assitant in the steps of the surgery in order to perform the surgery with less incisions and with the same safety
  Interventions: Procedure: Magnetic Gastric Bypass; Procedure: Magnetic Sleeve Gastrectomy; Procedure: Revisional Bariatric Surgery; Procedure: Nissen/Sleeve Gastrectomy with Magnetic Assistance; Procedure: Mangetic General Surgery

INTERVENTIONS:
Procedure: Magnetic Gastric Bypass — Perform a gastric bypass with the magnetic grasper to do the liver retraction, upper retraction of the stomach, upper retraction of the jejuno-jejunal anastomosis, upper retraction of the mesocolon to close petersen defect or the jejuno-jejunal anastomosis to close the intermesenteric defect also to do the retraction of the omega limb and perform the section of the limb and finish the gastric bypass
Procedure: Magnetic Sleeve Gastrectomy — Perform a sleeve gastrectomy with the magnetic grasper performing the liver retraction and the upper retraction of the stomach
Procedure: Revisional Bariatric Surgery — Perform liver retraction and also steps of the surgery like upper retraction of the stomach, upper retraction of the jejuno-jejunal anastomosis, upper retraction of the mesocolon to close petersen defect or the jejuno-jejunal anastomosis to close the intermesenteric defect also to do the retraction of the omega limb, upper retraction of the stomach
Procedure: Nissen/Sleeve Gastrectomy with Magnetic Assistance — Perform a nissen-sleeve gastrectomy with the magnetic grasper performing the liver retraction and the upper retraction of the stomach, retraction of the stomach to close the hiatal defect and perform a nissen funduplication before do the sleeve gastrectomy
Procedure: Mangetic General Surgery — Use the magnetic grasper to do the gallbladder retraction in cholecystectomies and upper retraction of the stomach to close the defect on hiatal hernia cases.

SUMMARY:
Magnetic devices have been successfully used in bariatric surgery. To the date the only reported use of the magnet was for liver retraction. This study is to demonstrate the safety and viability of using the magnetic system as a second surgical assistant in bariatric surgery and not only for liver retraction.

DETAILED DESCRIPTION:
Patients undergoing primary laparoscopic sleeve gastrectomy (SG), one-anastomosis gastric bypass (OAGB), and Roux-en-Y gastric bypass (RYGB) or revisional surgery by single-port or port-reduced approach.

Also others procedures like Nissen/Sleeve gastrectomy or general surgery. The magnetic system can be used like a second assistant in the steps of the surgery for example: liver retraction, upper retraction of gallbladder, retraction of the stomach, upper retraction of jejuno-jejunal anastomosis performing a gastric bypass or closing mesenteric defects liker intermesenteric or Petersen´s defect.

Using the single-port device or port-reduced approach to obtain better aesthetic results.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* BMI Greater than 30 kg/m2 (Obesity)
* Candidate to bariatric surgery
* GERD
* Candidate to revisional bariatric surgery
* Cholecystitis or Gallstones (General Surgery)

Exclusion Criteria:

* Patients with pacemakers or electromedical implants
* Uncontrolled metabolic diseases
* Psychiatric problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pantients candidates to bariatric surgery of the international unit of bariatric and metabolic surgery
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Rate of surgical complications | 1-2 hours
  Any complications or adverse event during the surgery
Range of surgical time | 1-2 hours
  See if the surgical time is kept normal
Rate of complications related to the magnetic system | 1-2
  Any adverse event or complication related to the magnetic system use during the surgery
Outcomes of magnetic grasper acting like a second assistant | 1-2 hours
  See if the magnetic system it can be used in any step of the surgery like a second surgical assistant

CONTACTS AND LOCATIONS:
Overall Officials: Andres Maldonado, MD, Principal Investigator — International Unit of Bariatric and Metabolic Surgery; Ali Urdaneta, MD. PhD., Principal Investigator — International Unit of Bariatric and Metabolic Surgery
Locations (1):
- Unidad Internacional de Cirugía Bariátrica y Metabólica, Maracaibo, Zulia, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided